CLINICAL TRIAL: NCT01191333
Title: CSP #556 - The Effectiveness of rTMS in Depressed VA Patients
Brief Title: The Effectiveness of rTMS in Depressed VA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 556
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Major Depressive Disorder
Keywords: Mood Disorder; Depression; stress disorder, post-traumatic; Depressive Disorder; Stress Disorders, Traumatic; substance related disorders; Transcranial Magnetic Stimulation, repetitive; transcranial magnetic stimulation; Veterans; mental health
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders; Depression; Stress Disorders, Post-Traumatic; Depressive Disorder; Stress Disorders, Traumatic; Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS (Experimental): Those receiving experimental treatment will receive 20 to 30 sessions of rTMS in blocks of 5 sessions. The treatment will be delivered by trained medical personnel.
  Interventions: Device: rTMS
- Sham rTMS (Placebo Comparator): Those receiving the sham rTMS will receive 20 to 30 sessions of sham rTMS in blocks of 5 sessions. The treatment will be delivered by trained medical personnel.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: rTMS — Repetitive Transcranial Magnetic Stimulation
  Arms: Active rTMS
Device: Sham Device — Placebo Device that simulates active rTMS treatment
  Arms: Sham rTMS

SUMMARY:
The purpose of this multi-site trial is to determine if repetitive Transcranial Magnetic Stimulation (rTMS) helps people with depression who have not been helped by medications or who have not been helped enough by medications.

DETAILED DESCRIPTION:
Major depression occurs in about 10% of American outpatients every year and of those, approximately 20% respond incompletely or not at all to trials of antidepressants, mood stabilizers, or psychotherapy (Kaplan and Sadock, 1996; Keller et al 1992; Thase, 2004). Treatment as usual for these cases of treatment resistant major depression (TRMD) frequently involves increased risks and increased side effects, such as those seen in monoamine oxidase inhibitors (MAOIs) and electroconvulsive therapy (ECT). New TRMD treatments are needed, preferably without major safety concerns or side effects as seen with aggressive polypharmacy or ECT.

Repetitive transcranial magnetic stimulation (rTMS) is a method of delivering brain stimulation without the seizures or risks associated with ECT, nor the potential side effects and risks of MAOI therapy. Systematic review and meta-analysis of the studies to date, which are typically of a small scale, appear to show a positive effect in TRMD (Martin et al. 2003). With a minimal side effect profile, and the rarity of untoward events and side-effects (Pascual-Leone et al. 1993; Wassermann 1997), safety concerns regarding the use of rTMS are considerably less than with ECT. Given this, rTMS has the potential to be a significant advance in care, if it were shown to be effective in TRMD in VA patients.

The trials of rTMS performed to date have not included participants with comorbid disorders, such as substance abuse and post-traumatic stress disorder (PTSD), thus the generalizability of their findings to a VA population is not clear. Further research including Veterans with possible comorbid disorders is necessary, given the high rates of co-occurring substance abuse and PTSD that is present in the Veteran population.

The present study is a randomized, controlled trial that compares active rTMS to a sham condition in Veterans with treatment resistant major depression and possible comorbid post-traumatic stress disorder (PTSD) and / or a history of substance abuse. Veterans will remain under the care of their VA primary mental health provider throughout the project. Participants will be assessed at pre-, mid- and several post-treatment time points. This is a multisite trial that will be conducted at 9 VA Medical Centers around the country.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 80 years of age
* Using the Structured Clinical Interview for Diagnostic and Statistical Manual (DSM) Disorders (SCID) for DSM-IV-TR (First et al. 2002) patients will be diagnosed Major Depressive Disorder (MDD).
* Have a Hamilton Rating Scale for Depression (HRSD-24) score greater or equal to 20 no more than 7 days prior to randomization.
* Exhibit moderate level of resistance to antidepressant treatment defined, using the Antidepressant Treatment History Form (ATHF) (Sackeim et al. 1990), as failure of at least two adequate medication trials.
* Duration of current episode of less than or equal to 10 years.
* Ability to obtain a Motor Threshold (MT) (should be determined at the end of the screening process).
* Currently under the care of a VA psychiatrist.
* If on a psychotropic medication regimen, that regimen will be stable for at least 4 weeks prior to randomization and patient will be willing to remain on a stable regimen during the acute treatment phase.
* Has an adequately stable condition and environment to enable attendance at scheduled clinic visits.
* For female participants, agrees to use one of the following acceptable methods of birth control

  * Complete abstinence (not having sexual intercourse with anyone)
  * An oral contraceptive (birth control pills)
  * Norplant
  * Depo-Provera
  * A condom with spermicide
  * A cervical cap with spermicide
  * A diaphragm with spermicide
  * An Intrauterine device
  * Surgical sterilization (having tubes tied)
* Able to read, verbalize understanding and voluntarily sign the Informed Consent Form prior to performance of any study-specific procedures or assessments.

Exclusion Criteria:

* Pregnant or lactating female (This is an FDA-required exclusion. In the future, if rTMS becomes a proven treatment for major depression, its safety in the context of pregnancy should be studied separately (Nahas et al. 1999).
* Unable to be safely withdrawn, at least two-weeks prior to treatment commencement, from medications that substantially increase the risk of having seizures. For the purpose of this study, those medications are listed in Appendix G (for example, theophylline).
* Have a cardiac pacemaker.
* Have an implanted device (deep brain stimulation) or metal in the brain.
* Have a cochlear implant.
* Have a mass lesion, cerebral infarct, increased intracranial pressure, or other active central nervous system (CNS) disease, including a seizure disorder.
* Known current psychosis as determined by DSM-IV or SCID (axis I, psychotic disorder, schizophrenia) or a history of a non-mood psychotic disorder.
* Known current Bipolar I disorder as determined by SCID or a History of Bipolar I disorder.
* Current amnestic disorders, dementia, Blessed Orientation-Memory-Concentration (BOMC) greater than 10, delirium, or other cognitive disorders.
* Current substance abuse (not including caffeine or nicotine) as determined by positive toxicology screen, or by history via SCID, within 3 months prior to screening.
* Patients with an elevated risk of seizure due to traumatic brain injury (TBI).
* Participation in another concurrent clinical trial.
* Patients with prior exposure to rTMS.
* Active current suicidal intent or plan as evidenced by a score of 4 or 5 on the suicidal ideation portion of the Columbia Suicide Severity Rating Scale (C-SSRS) or the endorsement of an actual attempt, interrupted attempt, or an aborted attempt in the past 6 months. All patients will be required to establish a written safety plan involving their primary psychiatrist and the treatment team before entering the clinical trial (See Section X.B.8).
* Unstable cardiac disease or recent (< 3 months previous) myocardial infarction.
* Patient refuses to sign consent for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2012-07-02 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome A. Yesavage, MD, Study Chair — VA Palo Alto Health Care System, Palo Alto, CA
Locations (9):
- United States (9):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Central Texas Veterans Health Care System, Temple, TX, Temple, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mi Z, Biswas K, Fairchild JK, Davis-Karim A, Phibbs CS, Forman SD, Thase M, Georgette G, Beale T, Pittman D, McNerney MW, Rosen A, Huang GD, George M, Noda A, Yesavage JA. Repetitive transcranial magnetic stimulation (rTMS) for treatment-resistant major depression (TRMD) Veteran patients: study protocol for a randomized controlled trial. Trials. 2017 Sep 2;18(1):409. doi: 10.1186/s13063-017-2125-y. PMID 28865495
- [Derived] Yesavage JA, Fairchild JK, Mi Z, Biswas K, Davis-Karim A, Phibbs CS, Forman SD, Thase M, Williams LM, Etkin A, O'Hara R, Georgette G, Beale T, Huang GD, Noda A, George MS; VA Cooperative Studies Program Study Team. Effect of Repetitive Transcranial Magnetic Stimulation on Treatment-Resistant Major Depression in US Veterans: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Sep 1;75(9):884-893. doi: 10.1001/jamapsychiatry.2018.1483. PMID 29955803

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 81 | 83
Completed | 60 | 65
Not Completed | 21 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 81 | 83 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (12.2) | 54.8 (12.6) | 55.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 67 | 65 | 132
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 14 | 26
  White | 63 | 63 | 126
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 81 | 83 | 164
Beck Scale for Suicide Ideation (BSI) [Mean (Standard Deviation); unit: units on a scale] — This self-report measure consists of 21 items with overall score range from 0 - 38, with the last two items not counted in scoring. A high score represents a worse outcome. Population: Missing values
  units on a scale
    number analyzed (Participants) | 77 | 82 | 159
    (all) | 3.7 (6.0) | 5.6 (6.7) | 4.7 (6.5)
Beck Depression Inventory (BDI) [Mean (Standard Deviation); unit: units on a scale] — This measure is a 21-item self-report test presented in a multiple choice format which measures presence and extent of depression with overall score range from 0 - 63. A higher score represents a worse outcome. Population: Missing values
  units on a scale
    number analyzed (Participants) | 78 | 77 | 155
    (all) | 22.6 (10.3) | 26.5 (10.0) | 24.5 (10.3)
VR-36 Mental Component Summary (MCS) [Mean (Standard Deviation); unit: units on a scale] — Standardized scoring ranging from 0-100. A higher score represents a better outcome Population: Missing value
  units on a scale
    number analyzed (Participants) | 81 | 82 | 163
    (all) | 27.2 (11.6) | 25.1 (10.0) | 26.2 (10.8)
VR-36 Physical Component Summary (PCS) [Mean (Standard Deviation); unit: units on a scale] — Standardized scoring ranging from 0-100. A higher score represents a better outcome Population: Missing value
  units on a scale
    number analyzed (Participants) | 81 | 82 | 163
    (all) | 42.4 (11.5) | 40.2 (10.0) | 41.3 (10.8)
Montgomery Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — As another measure of depression, the Montgomery-Asberg Depression Rating Scale (MADRS) has been used with increasing frequency in recent years to measure outcome in antidepressant efficacy trials. It offers an alternative view of depressive illness, and may be sensitive to depressive symptoms that are not easily captured in the context of the HRSD, such as hypersomnia, increased appetite, and concentration/indecision. The MADRS is a 10-item clinician rating of depressive symptoms. Each item is scored on a 7-point scale (0 to 6) (range 0-60).
  units on a scale | 24.7 (7.6) | 26.2 (6.9) | 25.5 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Achieving Remission From Depression as Assessed by Hamilton Rating Scale for Depression
Description: The primary outcome is a proportion of participants achieving remission from depression based on the HRSD24 less than or equal to 10 at the end of the acute treatment phase. 24 item Instrument with overall score range from 0 - 76. High values represent a worse outcome.
Time Frame: End of acute treatment 4-6 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 81 | 83
Participants | 33 | 31

2. Secondary Outcome: Mean Suicidal Ideation Score as Assessed by Beck Scale for Suicide Ideation (BSS)
Description: To help clinicians screen psychiatric patients for suicidal ideation, the Beck Scale for Suicide Ideation was developed, and is herein referred to as the BSS. This self-report measure consists of 21 items with overall score range from 0 - 38, with the last two items not counted in scoring. A high score represents a worse outcome.
Time Frame: End of acute treatment 4-6 weeks, then end of F/U 6 months
Population: ITT minus participants with missing values
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 67 | 72
units on a scale
  End of Acute Treatment | 2.0 (4.6) | 2.7 (4.9)
  End of F/U | 1.5 (4.2) | 2.5 (4.9)

3. Secondary Outcome: Mean Depression Score as Assessed by Beck Depression Inventory (BDI)
Description: This measure is a 21-item self-report test presented in a multiple choice format which measures presence and extent of depression with overall score range from 0 - 63. A higher score represents a worse outcome. Each of the 21 items addresses a specific symptom or attitude that pertains to depressed patients, and which are consistent with descriptions of the depression within the peer-reviewed literature. While generally deemed less reliable than scales score by a trained rater (for example, the HRSD), the Beck scale is easy to administer, and provides convenient means by which patients can effectively communicate their own perception of their mood state.
Time Frame: Baseline - end of acute treatment 4-6 weeks, then end of F/U 6 months
Population: ITT minus participants with missing values
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 66 | 72
units on a scale
  End of Acute Treatment | 14.2 (10.9) | 13.0 (9.5)
  End of F/U | 9.0 (8.3) | 12.8 (10.8)

4. Secondary Outcome: Mean Mental Component Score as Assessed by VR-36 Mental Component Summary (MCS)
Description: The VR-36 is a self-administered survey that measures eight dimensions of health: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. It yields scale scores for each of these eight health domains, and two summary measures of physical and mental health: the Physical Component Summary (PCS) and Mental Component Summary (MCS). MCS is analyzed in this section. Standardized scoring ranging from 0-100. A higher score represents a better outcome.
Time Frame: End of acute treatment 4-6 weeks, then end of F/U 6 months
Population: ITT minus participants with missing values
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 68 | 73
units on a scale
  End of Acute Treatment | 35.1 (14.3) | 36.0 (14.7)
  End of F/U | 34.5 (12.8) | 34.8 (13.4)

5. Secondary Outcome: Mean Physical Component Score as Assessed by VR-36 Physical Component Summary (PCS)
Description: The VR-36 is a self-administered survey that measures eight dimensions of health: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. It yields scale scores for each of these eight health domains, and two summary measures of physical and mental health: the Physical Component Summary (PCS) and Mental Component Summary (MCS). PCS is analyzed in this section. Standardized scoring ranging from 0-100. A higher score represents a better outcome.
Time Frame: End of acute treatment 4-6 weeks, then end of F/U 6 months
Population: ITT minus participants with missing values
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 68 | 73
units on a scale
  End of Acute Treatment | 41.9 (10.9) | 41.2 (11.9)
  End of F/U | 42.8 (10.8) | 40.1 (12.3)

6. Secondary Outcome: Mean Depression Score as Assessed by the Montgomery Asberg Depression Rating Scale (MADRS)
Description: As another measure of depression, the Montgomery-Asberg Depression Rating Scale (MADRS) has been used with increasing frequency in recent years to measure outcome in antidepressant efficacy trials. It offers an alternative view of depressive illness, and may be sensitive to depressive symptoms that are not easily captured in the context of the HRSD, such as hypersomnia, increased appetite, and concentration/indecision. The MADRS is a 10-item clinician rating of depressive symptoms. Each item is scored on a 7-point scale (0 to 6) (range 0-60). A high score represents a worse outcome.
Time Frame: End of acute treatment 4-6 weeks, then end of F/U 6 months
Population: ITT minus participants with missing values
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 70 | 74
units on a scale
  End of Acute Treatment | 14.3 (11.1) | 13.1 (10.5)
  End of F/U | 13.7 (10.2) | 15.0 (9.7)

ADVERSE EVENTS:
Time Frame: From informed consent until termination. 7-8 months.
Arm/Group | Active rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/83
Serious Adverse Events (participants affected / at risk) | 22/81 | 18/83
Other Adverse Events (participants affected / at risk) | 71/81 | 69/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (N=81) | Sham rTMS (N=83)
Suicidal ideation (Psychiatric disorders) | 4 (4) | 4 (4)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acoustic stimulation tests abnormal (Investigations) | 4 (4) | 5 (5)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (N=81) | Sham rTMS (N=83)
Nasopharyngitis (Infections and infestations) | 8 (8) | 8 (12)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (5)
Gastroenteritis (Infections and infestations) | 4 (5) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2) | 3 (3)
Influenza (Infections and infestations) | 1 (2) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 2 (3)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Tooth abscess (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Epididymitis (Infections and infestations) | 1 (2) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Vaginitis gardnerella (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 15 (25) | 16 (25)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Balance disorder (Nervous system disorders) | 0 (0) | 2 (2)
Sinus headache (Nervous system disorders) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Mononeuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Phantom pain (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acoustic stimulation tests abnormal (Investigations) | 16 (18) | 16 (19)
Colonoscopy (Investigations) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Protein total decreased (Investigations) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 6 (6)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ear canal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incorrect dosage administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Penis injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 6 (7) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Agitated depression (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Derealisation (Psychiatric disorders) | 1 (1) | 0 (0)
Dissociation (Psychiatric disorders) | 1 (1) | 0 (0)
Flashback (Psychiatric disorders) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Parasomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 3 (3) | 4 (4)
Adverse drug reaction (General disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Nodule (General disorders) | 0 (0) | 1 (1)
Sensation of blood flow (General disorders) | 0 (0) | 1 (1)
Sensation of foreign body (General disorders) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1)
Ulcer (General disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin discomfort (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 3 (3) | 0 (0)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Episcleritis (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 2 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 1 (1)
Dental care (Surgical and medical procedures) | 1 (1) | 0 (0)
Elective procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Papilloma excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 (3) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT01191333/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT01191333/SAP_001.pdf